CLINICAL TRIAL: NCT05933655
Title: Re-thinking the Role of Peers And Training Patients [RePeAT]
Acronym: RePeAT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Mechelle Sanders, Assistant Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 18638; K01HL159046 (NIH)
Record Dates: First submitted 2023-06-12; First posted 2023-07-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-06

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: . Patients will be randomized at a 1:1 ratio, stratified by the clinician.
Who Masked: Care Provider
Masking Description: Immediately after subjects complete the baseline surveys they will be randomized. The research coordinator will open a sealed envelope that specifies which group the subject is in. Neither the subject nor the research coordinator can choose the randomization group. The randomizations envelopes will be prepared
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peer Coach (Experimental): The research coordinator will set up a time for the subject to have a brief discussion with a peer coach from the study team approximately 1 week after randomization. During the coaching session, the peer coach will encourage the subject to mention their heart health goals to their primary care clinician during their next primary care appointment. The peer coach will also help the subject brainstorm ways to remove any barriers that may prevent them from having the discussion with their clinician. The peer coaching session and the subsequent medical appointment will be audio-recorded.
  Interventions: Behavioral: Peer Coach
- Control (No Intervention): The subject will not be asked to meet with the peer coach or anyone from the study team prior to their next visit with their primary care clinician. Their subsequent primary care appointment will be audio-recorded.

INTERVENTIONS:
Behavioral: Peer Coach — Peer coaching session to support shared decision making among patient with limited health literacy.
  Arms: Peer Coach

SUMMARY:
This study, Re-thinking the role of Peers And Training Patients [RePeAT], is designed to test the feasibility of training peer-coaches to prepare limited health literacy (LHL) patients to engage in shared-decision making (SDM) for cardiovascular disease (CVD) risk-reduction.

DETAILED DESCRIPTION:
The investigators will use a 2-arm pilot RCT design to assess the feasibility, and acceptability of the intervention. Up to 60 primary care patients will be randomly assigned to participate in the peer-coaching or control group. Patients will be randomized at a 1:1 ratio, stratified by the clinician. Half of the subjects (n=30) will be assigned to the peer-coaching intervention, and the other half will be assigned to the control group.

ELIGIBILITY:
Inclusion Criteria:

* A patient of Highland Family Medicine practice
* At least 40 years old and no more than 75 years old
* Be at ≥10% risk for CVD as calculated using the ASCVD Risk Estimator Plus
* No plans to leave the practice in the next 12 months
* English speaking
* Limited Health Literacy (self-report)

Exclusion Criteria:

* Have experienced a prior cardiac or vascular event such as myocardial infarction (MI) or cerebrovascular accident (CVA) or have had a CVD procedure such as installation of a stent or angioplasty
* Gave peripheral vascular disease, intermittent claudication or peripheral arterial disease
* Lack of capacity to consent

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2026-01-31 (Actual); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
ABCS Discussion | patient-clinician office visit, approximately 1 week after the peer coaching session
  The investigators will qualitatively code the office visit to determine if subjects engaged in a discussion with their clinician about their ABCS options/preferences.

SECONDARY OUTCOMES:
Peer Coach Fidelity | post-coaching, approximately 1-2 weeks prior to the patient-clinician office visit
  The investigators will qualitatively code the peer coaching sessions to determine if peer coaches used Teach-back during their session and if the coaching session was done with fidelity.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No